CLINICAL TRIAL: NCT03120741
Title: Dementia Patient's Behavior Evaluation Using Noninvasive Ambient Sensor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201608004RINB
Record Dates: First submitted 2016-11-15; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2016-12

CONDITIONS: Mild Cognitive Impairment, Dementia
Keywords: Healthcare Quality
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an observational study that uses daily activity and environmental sensing techniques to establish behavioral models of early dementia patients and cognitive healthy function to assess their daily behavior and determine their activities. Specifically, the team will collect information on a number of wireless sensors for dementia, mild cognitive impairment and healthy elderly residents, and use special mathematical models to establish the behavior of the two groups of subjects Model. The model will be developed a reliable algorithm to assess health risk of the subjects.

DETAILED DESCRIPTION:
With the help of intelligent home environment and Pervasive Computing, it is possible to bring information about the behavior of the patients to the caregivers and their relatives. In this study, non-invasive wireless sensors such as infrared motion sensor the switch sensor will be built in the home of the subjects. The wireless sensor data collected by the input to the team's "activity identification system" in order to assess the mathematical model of the subjects "capacity" and immediate judgment of their activities. In the identification of activities can be divided into two categories of behavior, risk behavior (harmful to the subjects) and protective behavior (beneficial to the subjects), real-time activity detection, can avoid dangerous behavior, such as water and gas off, roaming , Repetitive behavior (over-eating), forgetting to eat and day-night reversal (sleep disturbance), etc., the protection of behavior can be observed through a long time to help patients conduct beneficial behavior, such as regular quantitative diet.

ELIGIBILITY:
Inclusion criteria:

* Can communicate in Mandarin or Taiwanese.
* Consciousness is clear.
* Can do the daily activity by their own.

Exclusion criteria:

* Have a serious cardiopulmonary disease or physical activity is limited to those unable to carry out daily activities.
* Consciousness is not clear.
* Difficult communication, such as: aphasia patients, the use of respirator patients.
* Suffering from serious mental illness that can not match.
* Adopt absolute isolation, such as: open tuberculosis patients.
* Hearing or severe visual impairment that can not match.
* Can not exercise their consent.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The age of the subject is over 65. The education level is junior high school degree or above. The healthy elders will be selected by the MMSE score (over 24), AD-8 score (under 2) and the Mini-Cog (over 4).
  The MMSE score of the subjects with cognitive impairment or dementia is 10 to 23.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The relationship between moving pattern change and dementia. | 6 months
  Motion sensors will be installed on the ceiling. We will analyze multiple sensors to see how the participant move from one location to another. The data whether the participant is wandering or not and times of wandering will be measured.
The relationship between daily routine change and dementia. | 6 months
  Motion sensors, switch sensors, and current sensors will be installed in the home of the participant.
  The room which the participant is in, the appliance which the participant is using will be measured.
The relationship between sleeping time change and dementia. | 6 months
  Motion sensors will be installed in the bed or on the ceiling. The time when the participant goes to sleep, and the times the participant turns over during sleep will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chen Fu, Doctor, Principal Investigator — National Taiwan University, Department of Computer Science & Information Engineering
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan